CLINICAL TRIAL: NCT06842394
Title: Can Increased Medical Competence Reduce State Anxiety in Junior Doctors in the Emergency Department: a Randomized Controlled Trial
Brief Title: Can Increased Medical Competence Reduce State Anxiety in Junior Doctors in the Emergency Department?
Acronym: MINDED
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anna Sofie Mundt, Principal Investigator, Copenhagen Academy for Medical Education and Simulation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: F-24053546
Record Dates: First submitted 2025-02-06; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: State Anxiety; Psychological Stress; Education, Medical; E-learning; Acute Medical Unit
Keywords: Junior Doctors; Emergency Department; Adaptive E-learning; Medical Competence; Medical Education; Healthcare Workforce; state anxiety
MeSH Terms: conditions — Anxiety Disorders; Stress, Psychological; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adaptive e-learning (Experimental): The intervention group will receive the adaptive e-learning program in addition to standard onboarding within the first six weeks of employment
  Interventions: Other: Adaptive E-learning
- Standard onboarding (No Intervention): The control group will receive standard onboarding

INTERVENTIONS:
Other: Adaptive E-learning — An adaptive e-learning program comprising 13 modules each unfolding and testing the learners knowledge and ability to assess own competence regarding specific acute and time critical medical patient conditions.
  Arms: Adaptive e-learning

SUMMARY:
This randomized controlled trial investigates whether an adaptive e-learning program on acute and time critical medical conditions can reduce state anxiety and improve the competence of junior doctors working in emergency departments. Junior doctors assigned to frontline shifts will be enrolled and randomized into two groups: an intervention group receiving the e-learning program within the first six weeks of employment and a control group receiving standard onboarding with delayed access to the program. The primary outcome is the change in state anxiety levels, assessed using the State-Trait Anxiety Inventory (STAI-6). Secondary outcomes include perceived self-efficacy during shifts and self-assessed competency improvements.

DETAILED DESCRIPTION:
The healthcare system is under increasing pressure due to demographic changes, including a growing elderly population and a shrinking workforce. This intensifies the challenges of recruiting and retaining healthcare professionals, particularly in high-stress environments like emergency departments. Junior doctors often face significant anxiety during their early careers, which is associated with higher rates of burnout, decreased job satisfaction, and early career attrition Transitioning from medical education to clinical practice is a critical period marked by high levels of stress and anxiety. Research highlights that new doctors frequently report feeling inadequately prepared for the demands of clinical work, particularly in acute care settings where decision-making is both time-sensitive and impactful. Anxiety during this transition is not only detrimental to individual well-being but also impacts patient safety and care quality.

Prior interventions, including simulation-based training and e-learning programs, have shown promise in reducing stress and improving clinical competence among healthcare professionals. For example, adaptive e-learning platforms have demonstrated efficacy in tailoring content to individual learners' needs, enhancing knowledge retention, and fostering confidence in clinical skills.

Building on this evidence, the MINDED trial (MedIcal juNior Doctors Emergency Department) aims to evaluate the impact of an adaptive e-learning program tailored specifically for junior doctors in emergency medicine. This program is designed to improve their theoretical knowledge and practical competencies, thereby reducing anxiety and enhancing performance during emergency shifts. By addressing both psychological and educational needs, the trial seeks to contribute to a more resilient and competent workforce in acute care.

Objectives

1. Primary Objective: To assess the impact of the adaptive e-learning program on reducing state anxiety levels in junior doctors.
2. Secondary Objectives: To evaluate improvements in perceived self-efficacy during shifts and competency following the intervention.

Hypotheses

1. Participation in the adaptive e-learning program will significantly reduce state anxiety compared to controls.
2. The adaptive e-learning program will enhance both objective and subjective medical competence among participants.

ELIGIBILITY:
Inclusion Criteria:

* Junior residents in front- or middle-level shifts in emergency departments across the Capital Region of Denmark.
* Employed between January 1, 2025, and April 31, 2025.

Exclusion Criteria:

* Prior exposure to the adaptive e-learning program.
* Denying participation.

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in STAI scores | Immediately after the intervention
  A change in STAI-6 scores from baseline to 6 weeks post-intervention.

SECONDARY OUTCOMES:
Changes in perceived selfefficacy during shifts, measured through a structured survey. | Immediately after the intervention
  The participants report self assesment on how they experience their selfefficacy after the interventions has been completed
Qualitative insights from interviews with participants exploring factors influencing anxiety and competency. | Immediately after the intervention
  Individual interviews with participants in the intervention group
• E-learning -based exploratory outcomes, including learning curves, self-assessed competencies to objective competencies, e-learning implementation and user satisfaction. | Immediately after the intervention
  The e.learning system extratcs data on learning curves, self-assessed competencies to objective competencies, which is combined with a survey on e-learning implementation and user satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Jonas P Eiberg, PhD, Principal Investigator — Department of Vascular Surgery, The Heart Center, University Hospital of Copenhagen - Rigshospitalet and Copenhagen Academy for Medical Education and Simulation
Locations (1):
- Emergency Departments in the Capital Region of Denmark, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No
The aim of this study is to generate data on how an e-learning programme may or may not effect STAI on younger doctors in general. Thus, the individual focus is less important and will not be discussed with other researchers.

REFERENCES:
- [Background] Ristić, I., Runić-Ristić, M., Savić Tot, T., Tot, V., & Bajac, M. B. (2023). The Effects and Effectiveness of An Adaptive E-Learning System on The Learning Process and Performance of Students. International Journal of Cognitive Research in Science, Engineering and Education, 1, 77-92.
- [Background] Juul MV, Fast AT, Lassen AT, Laugesen S. Anxiety among medical students and junior doctors in Denmark. Dan Med J. 2022 Sep 29;69(11):A03220162. PMID 36331149
- [Background] Piso B, Nussbaumer-Streit B, Gartlehner G. [WHO Guidelines on Mental Health at Work]. Gesundheitswesen. 2024 Mar;86(3):216-219. doi: 10.1055/a-2249-5787. Epub 2024 Mar 12. German. PMID 38471514
- [Background] Stassen P, Westerman D. Novice Doctors in the Emergency Department: A Scoping Review. Cureus. 2022 Jun 23;14(6):e26245. doi: 10.7759/cureus.26245. eCollection 2022 Jun. PMID 35898382
- [Background] Skov RAC, Lawaetz J, Konge L, Resch TA, Aasvang EK, Meyhoff CS, Westerlin L, Jensen MK, Eiberg JP. Role-reversal simulation training to enhance performance and reduce stress of endovascular scrub nurses in the operating room. Curr Probl Surg. 2024 Oct;61(10):101577. doi: 10.1016/j.cpsurg.2024.101577. Epub 2024 Jul 31. No abstract available. PMID 39266129
- [Background] Shahsavari H, Ghiyasvandian S, Houser ML, Zakerimoghadam M, Kermanshahi SSN, Torabi S. Effect of a clinical skills refresher course on the clinical performance, anxiety and self-efficacy of the final year undergraduate nursing students. Nurse Educ Pract. 2017 Nov;27:151-156. doi: 10.1016/j.nepr.2017.08.006. Epub 2017 Aug 8. PMID 28910662
- [Background] Seathu Raman SS, McDonnell A, Beck M. Hospital doctor turnover and retention: a systematic review and new research pathway. J Health Organ Manag. 2024 Feb 27;38(9):45-71. doi: 10.1108/JHOM-04-2023-0129. PMID 38448230
- [Background] Saffari M, Bashar FR, Vahedian-Azimi A, Pourhoseingholi MA, Karimi L, Shamsizadeh M, Gohari-Moghadam K, Sahebkar A. Effect of a Multistage Educational Skill-Based Program on Nurse's Stress and Anxiety in the Intensive Care Setting: A Randomized Controlled Trial. Behav Neurol. 2021 Apr 26;2021:8811347. doi: 10.1155/2021/8811347. eCollection 2021. PMID 33986878
- [Background] Montgomery A, Panagopoulou E, Esmail A, Richards T, Maslach C. Burnout in healthcare: the case for organisational change. BMJ. 2019 Jul 30;366:l4774. doi: 10.1136/bmj.l4774. No abstract available. PMID 31362957
- [Background] Monrouxe LV, Bullock A, Gormley G, Kaufhold K, Kelly N, Roberts CE, Mattick K, Rees C. New graduate doctors' preparedness for practice: a multistakeholder, multicentre narrative study. BMJ Open. 2018 Aug 29;8(8):e023146. doi: 10.1136/bmjopen-2018-023146. PMID 30158236
- [Background] Mathisen J, Nguyen TL, Jense JH, Rugulies R, Rod NH. Reducing employee turnover in hospitals: estimating the effects of hypothetical improvements in the psychosocial work environment. Scand J Work Environ Health. 2021 Sep 1;47(6):456-465. doi: 10.5271/sjweh.3969. Epub 2021 May 30. PMID 34052852
- [Background] Klitgaard TL, Stentoft D, Skipper M, Gronkjaer M, Nohr SB. Struggling to fit the white coat and the role of contextual factors within a hospital organisation - an ethnographic study on the first months as newly graduated doctors. BMC Med Educ. 2021 Jan 25;21(1):74. doi: 10.1186/s12909-021-02493-2. PMID 33494741
- [Background] Fuster V. Changing Demographics: A New Approach to Global Health Care Due to the Aging Population. J Am Coll Cardiol. 2017 Jun 20;69(24):3002-3005. doi: 10.1016/j.jacc.2017.05.013. No abstract available. PMID 28619199